CLINICAL TRIAL: NCT00236743
Title: Topiramate (RWJ 17021-000) Clinical Trial In Children With Partial Onset Seizures
Brief Title: A Study of the Effectiveness and Safety of Topiramate in the Treatment of Children With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005467
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy; Epilepsies, Partial; Seizures
Keywords: topiramate; epilepsy; partial epilepsies; partial epilepsy; seizures; epileptic seizures; partial seizure disorder; children; pediatric
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of oral topiramate as add-on therapy in children with uncontrolled partial onset seizures who are taking one or two standard anti-epileptic drugs.

DETAILED DESCRIPTION:
Epilepsy is characterized by seizures, which are abnormal electrical discharges in the brain that temporarily disrupt normal brain function. Seizures are classified as "generalized," originating in both sides of the brain simultaneously, or "partial-onset," starting in one area of the brain. Antiepilepsy medications, such as topiramate, are selected based on seizure type. This is a double-blind, placebo-controlled study that includes a baseline phase and a treatment phase. During the baseline phase (8 weeks duration), patients receive a stable dose of one or two standard antiepileptic drugs (AEDs), and the parent or guardian records the occurrences of seizure in a diary. Patients who continue to have seizures during treatment with standard AEDs proceed into the double-blind treatment phase. Patients then receive topiramate or placebo once daily at a dosage of 25 milligrams[mg] or 50 mg based on body weight (to 6mg/kg per day), increasing gradually to twice daily dosing at a maximum of 125-400 mg (based on body weight) for 112 days (16 weeks total duration of the double-blind phase), while continuing on their standard AED regimen. Assessments of effectiveness include the percent reduction in the average monthly seizure rate, percent of patients responding to treatment (having equal to or greater than 50% reduction in seizure rate), and the parent's or guardian's global assessment of medication at end of study. Safety assessments include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, chemistry, urinalysis), neurologic examinations, and vital sign measurements (blood pressure, pulse, body weight) at specific intervals during the treatment phase. The study hypothesis is that topiramate, taken as add-on therapy to treatment with AEDs, will significantly reduce seizure frequency, compared with placebo, in children with refractory partial epilepsy: that is, children who continue to have seizures despite treatment with first-line AEDs. In addition, it is hypothesized that topiramate is well-tolerated. Oral topiramate, daily for 112 days. Starting dose is 25 mg or 50mg, based on body weight. Maximum doses based on patient weight: 125 mg/day (36-54 pounds[lb]); 175 mg/day (55-74 lb); 225 mg/day (75-94 lb); and 400 mg/day (95 or more pounds). Matching placebo was used to maintain blinding.

ELIGIBILITY:
Inclusion Criteria:

* Patients must weigh at least 36 pounds (16 kilograms)
* patients must have partial onset seizures (with or without secondarily generalized seizures) being treated with at least one, but no more than two antiepileptic drugs (AEDs)
* patients must have at least 6 partial onset seizures during the 8-week baseline phase, with at least one seizure during each 4-week period
* an electroencephalogram (EEG) with features consistent with partial epilepsy performed prior to study initiation or during the baseline phase

Exclusion Criteria:

* Females who are pregnant, nursing, or those not using adequate birth control if capable of having children
* patients with a treatable cause of seizures (for example, infections)
* patients with a progressive disorder of the nervous system
* patients with a clinical diagnosis of Lennox-Gastaut syndrome
* patients with a history of generalized status epilepticus (repeated or prolonged seizures) while on appropriate anti-epileptic therapy

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 1994-06; Study Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the average monthly seizure rate from baseline to end of treatment

SECONDARY OUTCOMES:
Percent of patients responding to treatment (>= 50% reduction in seizure rate from baseline to end of treatment); parent's or guardian's global assessments at beginning of treatment and end of study; incidence of adverse events throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Ritter F, Glauser TA, Elterman RD, Wyllie E. Effectiveness, tolerability, and safety of topiramate in children with partial-onset seizures. Topiramate YP Study Group. Epilepsia. 2000;41(S1):82-5. doi: 10.1111/j.1528-1157.2000.tb02178.x. PMID 10768307
- See also: A study of the effectiveness and safety of topiramate in the treatment of children with epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=648&filename=CR005467_CSR.pdf